CLINICAL TRIAL: NCT03762083
Title: An Open-label Study to Evaluate Clinical Performance of Gedea Pessary in Adult Women With Bacterial Vaginosis
Brief Title: Clinical Performance of a Vaginal Pessary (pHyph) in Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QRS-CL2-003
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Bacterial Vaginosis
Keywords: vaginitis; vaginal disease; vulvovaginitis; genital disease, female; vaginitis, bacterial
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis; Vaginal Diseases; Vulvovaginitis; Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pHyph, Gedea Pessary (Experimental): Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of BV.
  Interventions: Device: pHyph generation I

INTERVENTIONS:
Device: pHyph generation I — A vaginal tablet for the treatment of BV with administration every 48 hours.
  Other Names: Gedea pessary

SUMMARY:
This is an open-label, single-armed, multi-center study to evaluate clinical performance, tolerability, and safety of Gedea Pessary in 24 adult women with confirmed bacterial vaginosis (BV) according to fulfillment of at least 3 of the 4 Amsel criteria. On Day 0, patients will have gynecological examination, vaginal samples taken, and will receive the investigational product to be self-administered. Patients will be examined after 7 days with respect to 3 Amsel criteria (the criterion: "pH of vaginal fluid above 4.5" is only included at study inclusion for diagnosis), and if not cured, will receive prolonged treatment for one additional week. Patients will be followed-up by telephone up to 29 days after last treatment. Vaginal samples will be used for confirming diagnosis and microbiome analyzes. Patient questionnaires will be used for assessing BV symptoms, usability, and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

Adult, post-menarchal, pre-menopausal women aged 18 years or older

* Diagnosis of BV according to Amsel's criteria, defined as having at least 3 of the 4 following criteria:

  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (more than 20 percent of epithelial cells)
  3. pH of vaginal fluid above 4.5
  4. Release of fishy odor "i.e. a positive whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added
* Having decisional capacity and providing written informed consent
* Negative urine pregnancy test at screening
* Refrain from using any intravaginal products (i.e., contraceptive creams, gels, foams, sponges, lubricants, or tampons, etc.) during the study period
* Refrain from sexual intercourse or use a condom until Day 7
* Signed informed consent and willing and able to comply with all study requirements

Exclusion Criteria:

Patients with known or apparent signs of other infectious causes of BV (vulvovaginal candidiasis, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at screening

* Anticipated menstruation during the treatment period (Day 0 till Day 7)
* Patients who are pregnant or breastfeeding
* Patients who were treated for BV within the past 14 days
* Patients who are currently receiving antibiotic therapy unrelated to BV or have received antibiotic therapy within the past 14 days
* Patients who have used pH-modifying vaginal products within the last 14 days
* Patients who have received an investigational drug in a clinical investigation within 30 days prior to screening
* Known/previous allergy or hypersensitivity to any product constituent
* Any medical condition that in the Investigator's judgments would make the patient unsuitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Cardell, MD, PhD, Principal Investigator — Kvinnokliniken, Region Skåne
Locations (2):
- Sweden (2):
  - Stortorgets Gynekologmottagning, Helsingborg
  - Sophiakliniken, Lund

REFERENCES:
- See also: Sponsor webpage — http://gedeabiotech.com

RESULTS

PARTICIPANT FLOW:
Groups:
- pHyph, Gedea Pessary: Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of bacterial vaginosis (BV).
  pHyph, Gedea pessary: pHyph is a vaginal tablet for the treatment of BV.
Period: Overall Study
Arm/Group | pHyph, Gedea Pessary
Started | 24 (Received study treatment.)
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: A total of 24 participants were enrolled, and all 24 participants received study treatment.
Groups:
- pHyph, Gedea Pessary: Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of BV.
  pHyph, Gedea pessary: pHyph is a vaginal tablet for the treatment of BV.
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 24
Experience any bacterial vaginosis (BV) infection during the last 12 months [Count of Participants; unit: Participants]
  Yes | 16
  No | 8

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: Defined as absence of all of the following 3 Amsel criteria:
  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (more than 20% of epithelial cells)
  3. Release of fishy odor "i.e. a positive whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added
Time Frame: Day 7
Population: Number of patients included in analysis = 22.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Participants | 18
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; It was assumed that the true cure rate was equal to 70%, therefore 22 patients were needed to obtain 90% chance (90% power) to show that the one-sided 95% confidence interval (CI) for the observed cure rate was above 40%. Hypotheses for the primary clinical performance endpoint: * Null hypothesis: Clinical cure rate is less than or equal to 40%. * Alternative hypothesis (one-sided): Clinical cure rate is above 40%; Test type: Other — The clinical performance endpoint - Clinical cure rate on Day 7 - was calculated and presented together with a one-sided 95% CI based on the exact binomial distribution (Clopper-Pearson); Clinical cure rate = 81.9, 95% CI 1-sided [lower limit 63.1]

2. Secondary Outcome: Proportion of Patients Being Negative for Each of the 3 Amsel Criteria - Criterion 1
Description: Defined as absence of one of the following Amsel criteria:
  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (more than 20% of epithelial cells)
  3. Release of fishy odor "i.e. a positive whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added
Time Frame: Day 7 compared to Day 0
Population: Statistical analysis of proportion of patients being negative for Amsel criterion 1 (discharge) on Day 7 compared to Day 0. Number of patients included in analysis =21.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 21
Participants | 18
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Prop. negative for Amsel criterion 1. = 85.7, 95% CI 2-sided [63.7 to 97.0]

3. Secondary Outcome: Proportion of Patients Being Negative for Each of the 3 Amsel Criteria - Criterion 2
Description: Defined as absence of one of the following Amsel criteria:
  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (more than 20% of epithelial cells)
  3. Release of fishy odor "i.e. a positive whiff test" when alkali (10% potassium hydroxide [KOH] solution is added
Time Frame: Day 7 compared to Day 0
Population: Statistical analysis of proportion of patients being negative for Amsel criterion 2 (clue cells) on Day 7 compared to Day 0. Number of patients included in analysis = 20.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 20
Participants | 18
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Prop. negative for Amsel criterion 2. = 90.0, 95% CI 2-sided [68.3 to 98.8]

4. Secondary Outcome: Proportion of Patients Being Negative for Each of the 3 Amsel Criteria - Criterion 3
Description: Defined as absence of one of the following Amsel criteria:
  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (more than 20% of epithelial cells)
  3. Release of fishy odour "i.e. a positive whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added
Time Frame: Day 7 compared to Day 0
Population: Statistical analysis of proportion of patients being negative for Amsel criterion 3 (fishy odour) on Day 7 compared to Day 0. Number of participants included in the analysis = 22.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Participants | 19
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Prop. negative for Amsel criterion 3. = 86.4, 95% CI 2-sided [65.1 to 97.1]

5. Secondary Outcome: Usability, Measured by Patient Questionnaire
Description: General assessment of the treatment on a integer scale that ranges from 1 to 10. The lower end of the scale is indicated with the term "Not satisfied" and the higher end with the term "Very satisfied".
  Question asked: How do you generally regard the treatment?
Time Frame: Day 7
Population: The Full analysis set population contained 24 patients. 2 patients were not included in this analysis due to missing data.
Measure: Mean (Standard Deviation); unit: Integer scale (1-10)
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Integer scale (1-10) | 7.1 (2.3)

6. Secondary Outcome: Proportion of Patients Having a Recurrence of the BV
Description: Proportion of patients answering Yes to the question "Have the symptoms recurred?"
Time Frame: Up to Day 35
Population: The Full analysis set population contained 24 patients.The sub-set of the Full analysis set including patients not receiving prolonged treatment contained 18 patients. Of these, 18 patients were included in this analysis of recurrence at Day 14 and 16 patients were included in the analysis of recurrence at Day 35.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 18
Participants
  Day 14 | 1
  Day 35: number analyzed (Participants) | 16
  Day 35 | 0
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Recurrence rate Day 14 = 5.6, 95% CI 2-sided [0.1 to 27.3]
Statistical Analysis 2: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Recurrence rate Day 35 = 0, 95% CI 2-sided [0 to 20.6]

ADVERSE EVENTS:
Time Frame: Up to day 42.
Arm/Group | pHyph, Gedea Pessary
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 11/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pHyph, Gedea Pessary (N=24)
Headache (Nervous system disorders) | 10 (13)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03762083/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03762083/SAP_001.pdf